CLINICAL TRIAL: NCT06401941
Title: The Impact of Staying in Hyperbaric Oxygen Conditions on the Oxidant-antioxidant Balance and the Activities of Selected Lysosomal Enzymes
Brief Title: Selected Lysosomal Enzyme Activities and the Oxidant-antioxidant Balance in Hyperbaric Oxygen Condition.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Paweł Sutkowy, PhD, Assistant professor, Nicolaus Copernicus University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KB 260/2016
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Hyperbaric Oxygenation; Oxygen Toxicity; Antioxidants; Oxidative Stress
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Hyperbaric oxygen (HBO) therapy.
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Controls (No Intervention): Healthy individuals that never treated with HBO therapy.

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — HBO session includes three 20-minute inhalations of pure oxygen in a hyperbaric chamber utilizing specially fitted face masks for each patient. The session is conducted as follows: 10 minutes compression of up to 2.5 atm (0.25 MPa), inhalation of 100% oxygen for 20 minutes, a 5-minute break in the chamber without the mask (oxygen concentration up to 23%, constant temperature (room) and humidity), again 20 minutes inhalation of 100% oxygen, another 5-minute break (the same condition), the last 20 minutes inhalation of 100% oxygen, and finally a 10-minute decompression. The total duration of the session was 90 minutes.
  Other Names: HBO treatment; Hyperbaric Oxygenation
  Arms: Patients

SUMMARY:
The aim of the research project was to investigate the effects of hyperbaric oxygen (HBO) treatment on the redox equilibrium in individuals with different pathological conditions. Both hyperbaric oxygenation and the pathological condition are associated with redox imbalance (oxidative stress), however, HBO is successfully used in the treatment of chronic wounds, e.g., diabetic foot syndrome, as well as in sudden and acute hearing loss, e.g., acute acoustic trauma or idiopathic sudden sensorineural hearing loss.

DETAILED DESCRIPTION:
The study involed in sudden sensorineural hearing loss (SSNHL) patients, individuals with difficult-to-heal skin wounds following mechanical injuries, and diabetic foot patients. HBO therapy, which involved inhalation of 100% oxygen at a pressure of 2.5 atm, consisted of 14-30 sessions depending on the clinical case. The study material was venous blood drawn three times: before and after the first session, and after the last HBO procedure. The following variables were evaluated: the concentrations of thiobarbituric acid reactive substances (TBARS), malondialdehyde (MDA) and conjugated dienes (CD) in plasma and erythrocytes, the activities of catalase (CAT), superoxide dismutase (SOD) and glutathione peroxidase (GPx) in erythrocytes, as well as, blood counts.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form for participation in the study

Exclusion Criteria:

* other pathological conditions (disorders, wounds, diseases)
* bad feeling of the participant on the day of the study,
* refraining from smoking, drinking alcohol, and the consumption of any dietary supplements that can affect the oxidant-antioxidant balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Thiobarbituric acid reactive substances (TBARS) | Three days, three different condition measurements
  Lipid peroxidation index represented by malondialdehyde (MDA), determined in plasma and erythrocytes.
Malondialdehyde (MDA) | Three days, three different condition measurements
  Lipid peroxidation index; pure MDA determined using high-performance liquid chromatography in plasma and erythrocytes.
Conjugated dienes (CD) | Three days, three different condition measurements
  Lipid peroxidation index, determined in plasma and erythrocytes.
Catalase (CAT) | Three days, three different condition measurements
  Antioxidant enzyme, determined in erythrocytes.
Superoxide dismutase (SOD) | Three days, three different condition measurements
  Antioxidant enzyme, determined in erythrocytes.
Glutathione peroxidase (GPx) | Three days, three different condition measurements
  Antioxidant enzyme, determined in erythrocytes.

SECONDARY OUTCOMES:
White blood cell count (WBC) | Two days, two different condition measurements
  Leukocytes found in peripheral blood with specyfication of their types: lymphocytes, monocytes, neutrophils, eosinophils, basophils.
Red blood cell count (RBS) | Two days, two different condition measurements
  Erythrocytes found in peripheral blood.
Hemoglobin (HGB) | Two days, two different condition measurements
  Mean concentration of hemoglobin in the blood.
Hematocrit (HCT) | Two days, two different condition measurements
  The percentage of red blood cells in the blood.
Mean corpuscular volume (MCV) | Two days, two different condition measurements
  Mean volume of erythrocytes in the blood.
Mean corpuscular hemoglobin (MCH) | Two days, two different condition measurements
  Mean mass of hemoglobin in an erythrocyte.
Mean corpuscular hemoglobin concentration (MCHC) | Two days, two different condition measurements
  MCH expressed in a unit of blood volume.
Red cell distribution width (RDW) | Two days, two different condition measurements
  Differences in the volume and size of erythrocytes.
Platelets (PLT) | Two days, two different condition measurements
  Thrombocytes found in peripheral blood.
Plateletcrit (PCT) | Two days, two different condition measurements
  Volume occupied by platelets in the blood.
Mean platelet volume (MPV) | Two days, two different condition measurements
  Mean volume of thrombocytes in the blood.
Platelet distribution width (PDW) | Two days, two different condition measurements
  Measurement of platelet anisocytosis calculated from the distribution of individual platelet volumes.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Sutkowy, PhD, Principal Investigator — Department of Medical Biology and Biochemistry, Ludwik Rydygier Collegium Medicum in Bydgoszcz, Nicolaus Copernicus University in Torun, Karlowicza 24, 85-092 Bydgoszcz, Poland
Locations (1):
- Department of Medical Biology and Biochemistry, Ludwik Rydygier Collegium Medicum in Bydgoszcz, Nicolaus Copernicus University in Torun, Karlowicza 24, 85-092 Bydgoszcz, Poland, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
There is no individual participant data (IPD) sharing plan.

REFERENCES:
- [Derived] Sutkowy P, Paprocki J, Piechocki J, Wozniak A. The impact of hyperbaric oxygen therapy on the redox balance of patients with diabetic foot syndrome. Free Radic Res. 2024 Nov;58(11):723-732. doi: 10.1080/10715762.2024.2417286. Epub 2024 Oct 19. PMID 39425927